CLINICAL TRIAL: NCT00498563
Title: Investigation to Determine the Effects of Mild Hypobaric Hypoxia on Sleep and Post-Sleep Neurobehavioral Performance
Brief Title: Effects of Mild Hypobaric Hypoxia on Sleep and Post-sleep Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Collaborators: The Boeing Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB#2006024
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Altitude; Hypoxia; Environmental Sleep Disorder
Keywords: high altitude; sleep; altitude illness; neurobehavioral manifestations; psychomotor performance; mood states
MeSH Terms: conditions — Hypoxia; Dyssomnias; Altitude Sickness; Neurobehavioral Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: altitude exposure in hypobaric chamber

SUMMARY:
Hypobaric hypoxia (decreased oxygen supply to body tissues due to low atmospheric pressure) caused by exposure to high altitude disrupts sleep. Sleep deprivation is associated with degraded post-sleep performance of neurobehavioral tasks. The lowest altitude at which sleep and/or post-sleep performance are affected is not known. The study hypothesis is that sleep and/or post-sleep performance of neurobehavioral tasks will occur due to hypobaric hypoxia at altitudes of 8,000 or less.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* age 30 to 60 years

Exclusion Criteria:

* sleep disorders or abnormal sleep patterns
* mood or psychiatric disorders including claustrophobia
* altitude exposure above 5,000 ft in the previous 2 months
* born or raised at terrestrial altitude 5,000 ft or greater
* conditions that would disqualify for FAA Medical Certificate
* acute medical conditions

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2006-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Quality and quantity of sleep measured by actigraphy and polysomnography Neurobehavioral performance measured by Psychomotor Vigilance Test (PVT) and Automated Neurophysiologic Assessment Metrics Battery (ANAM) | 7 hours; 4 hours

SECONDARY OUTCOMES:
Mood State measured by Profile of Mood States (POMS) Symptoms of altitude illness measured by Environmental Symptoms Questionnaire (ESQ IV) and Lake Louise Symptom Scores (LLS) | 20 hours

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Muhm, M.D., M.P.H., Principal Investigator — The Boeing Company; Paul B Rock, DO, PhD, Principal Investigator — Oklahoma State University Center for Aerospace & Hyperbaric Medicine
Locations (1):
- Oklahoma State University Center for Aerospace & Hyperbaric Medicine, Tulsa, Oklahoma, United States